CLINICAL TRIAL: NCT01181973
Title: An Open-label, Randomized, Phase 1, Single-Dose Crossover Study to Evaluate Safety, Tolerability and Relative Bioavailability of Pegvisomant 1 X 30 Mg Vs 2 X 15 Mg Subcutaneously Administered in Healthy Subjects
Brief Title: Safety, Tolerability and Relative Bioavailability of Pegvisomant in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A6291026
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Bioavailability
Keywords: Relative bioavailability; pegvisomant
MeSH Terms: interventions — pegvisomant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment sequence #1 (Active Comparator): One 1-mL subcutaneous injection at 30 mg/mL in Period 1 and two 1-mL subcutaneous injections at 15 mg/mL each in Period 2
  Interventions: Drug: pegvisomant
- Treatment sequence #2 (Active Comparator): Two 1-mL subcutaneous injections at 15 mg/mL each in Period 1 and one 1-mL SC injection at 30 mg/mL in Period 2
  Interventions: Drug: pegvisomant

INTERVENTIONS:
Drug: pegvisomant — One 1-mL subcutaneous injection at 30 mg/mL. A 30-mg vial is supplied as lyophilized powder. Each vial should be reconstituted with 1 mL of Sterile Water for Injection (WFI).
  Other Names: B2036-PEG
  Arms: Treatment sequence #1
Drug: pegvisomant — Two 1-mL subcutaneous injections at 15 mg/mL each. Two 15-mg vials are supplied as lyophilized powder. Each vial should be reconstituted with 1 mL of Sterile Water for Injection (WFI).
  Other Names: B2036-PEG
  Arms: Treatment sequence #1
Drug: pegvisomant — Two 1-mL subcutaneous injections at 15 mg/mL each. Two 15-mg vials are supplied as lyophilized powder. Each vial should be reconstituted with 1 mL of Sterile Water for Injection (WFI).
  Other Names: B2036-PEG
  Arms: Treatment sequence #2
Drug: pegvisomant — One 1-mL subcutaneous injection at 30 mg/mL. A 30-mg vial is supplied as lyophilized powder. Each vial should be reconstituted with 1 mL of Sterile Water for Injection (WFI).
  Other Names: B2036-PEG
  Arms: Treatment sequence #2

SUMMARY:
The hypothesis to be tested is that the bioavailability of the new 30-mg vial is similar to that of the current approved 15 -mg vials. In addition, the SC injection using the new 30-mg vial is safe and well-tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females between the ages of 21 and 55 years

Exclusion Criteria:

* Positive urine drug screen
* Excessive use of alcohol or nicotine-containing products
* Pregnant or nursing females

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The area under the pegvisomant concentration-time curve from time 0 to infinity hours post dose (AUCinf) | 16 days
The area under the pegvisomant concentration-time curve from time 0 to last observed timepoint (AUClast) | 16 days

SECONDARY OUTCOMES:
Maximal pegvisomant concentration (Cmax) | 16 days
The timepoint at which Cmax is obtained (Tmax) | 16 days
Elimination half-life of pegvisomant (as data permit) | 16 days
Biomarkers IGF-1 (A few samples will be taken at timepoints around Tmax to observe the pegvisomant effect on IGF-1) | 16 days
Safety laboratory tests (including hematology and serum chemistry parameters) and adverse events (including local site reactions) | 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6291026&StudyName=Safety%2C%20Tolerability%20and%20Relative%20Bioavailability%20of%20Pegvisomant%20in%20Healthy%20Subjects%20